CLINICAL TRIAL: NCT03972787
Title: Effects of a Proactive Social Robot for Older Adults in Reducing Loneliness and Social Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Collaborators: Jewish Senior Living Group (Unknown); Intuition Robotics (Unknown)
Responsible Party: Principal Investigator, Dr. Allison B. Sekuler, Sandra A Rotman Chair in Cognitive Neuroscience; Managing Director and Senior Scientist, Rotman Research Institute; Managing Director, Centre for Aging + Brain Health Innovation; Vice-President Research, Baycrest Health Sciences, Baycrest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB #18-54
Record Dates: First submitted 2019-05-24; First posted 2019-06-04 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Loneliness; Mood; Quality of Life

STUDY DESIGN:
Intervention Model Description: This study is a stratified, parallel, randomized waitlist control study that will be implemented at Baycrest and JSLG/UCSF, in which eligible, consented participants will be randomly allocated to the ElliQ (intervention) group or the waitlist control group following a 1:1 allocation ratio. In light of the potential benefits of ElliQ exposure, the waitlist control group will receive the ElliQ intervention after serving as a comparable contemporary control group for the ElliQ intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive Social Robot (Intervention) (Experimental): Participants will have the opportunity to use ElliQ for a total of 8 weeks to determine the impacts of the system on participants' loneliness, mood, technology use, and quality of life.
  Interventions: Device: Proactive social robot
- Waitlist Control (No Intervention): Participants will not receive any intervention for a total of 8 weeks to determine whether any impacts noted for participants' loneliness, mood, technology use, and quality of life are unique to ElliQ or are influenced by other factors.

INTERVENTIONS:
Device: Proactive social robot — ElliQ, is a new type of robotic technology aimed at reducing loneliness and social isolation in older adults. It differs from other social/companion robots on the market, as it leverages artificial intelligence to create personalized and interactive experiences for the user, while also proactively offering prompts (such as reminding the user to stay hydrated) and suggesting and initiating various activities for the user (such as offering to play a game). This social companion adapts to the personalities and interests of the older adult, creating a personalized experience and recommending content the user may enjoy such as news, music, TED talks, and cognitive games.
  Other Names: ElliQ
  Arms: Proactive Social Robot (Intervention)

SUMMARY:
This project will to evaluate whether a proactive social robot (ElliQ) has an impact on reducing social isolation and loneliness in older adults who are living alone, while also promoting independence and aging in place. To achieve this, the following research questions will be investigated:

1. How does the use of ElliQ impact the following outcomes in older adults:

   * Loneliness and social isolation;
   * Accessibility to and use of technology;
   * Quality of life, mood, and overall well-being; and
   * Caregiver experience?
2. Do particular characteristics of the older adult population influence these impacts?

DETAILED DESCRIPTION:
Study Design

Users

This study is a stratified, parallel, randomized waitlist control study that will be implemented at Baycrest and the Jewish Senior Living Group (JSLG), in which eligible, consented participants will be randomly allocated to the ElliQ (intervention) group or the waitlist control group following a 1:1 allocation ratio. In light of the potential benefits of ElliQ exposure, the waitlist control group will receive the ElliQ intervention after serving as a comparable contemporary control group for the ElliQ intervention group.

Those in the intervention group will first undergo participant characterization and baseline data collection (time 1; week 0). Shortly after, they will be provided with the ElliQ technology in their homes. They will then trial the device for 8 weeks (weeks 1-8). The 8-week trial will be followed with a post-trial data-collection session (time 2; week 9), where they will be asked to return the ElliQ system. At this time, participants will be asked to complete some of the same measures they completed at time 1, and they will also have the opportunity to take part in a one-time, audio-recorded focus group or interview, where field notes will be taken. Following this, the participants will not have a device from weeks 10-17; on week 18, they will be asked to attend a follow-up session (time 3; week 18), where they will be asked to complete some of the same measures they completed at times 1 and 2.

Those who get assigned to the second (waitlist) condition will attend an initial baseline data-collection session (time 1; week 0), where questionnaires related to participant characteristics and baseline measures will be administered. Participants will then wait for 8 weeks to get the ElliQ device (weeks 1-8). After this 8-week wait, participants will be invited to attend another data-collection session (time 2; week 9), where they will be asked to complete some of the same measures that they completed at time 1. Following this session, participants will trial the device for 8 weeks (weeks 10-17). After the 8-week trial, participants will be asked to attend a post-trial data-collection session (time 3; week 18), where they will return the ElliQ system. Participants will then complete a number of the same measures that were completed at times 1 and 2, and attend a one-time, audio-recorded focus group or interview session, where field notes will be taken.

Upon completion of the study tasks (i.e., at the final data-collection session at week 18), each participant's study participation will conclude.

Informal Caregivers

Informal caregivers (e.g., family, friends who provide care for the ElliQ user) may also be enrolled in the study to investigate their experiences with the messaging function of the ElliQ system (user and caregiver pairs will be referred to as "dyads" going forward). Of note, users who do not have caregivers can still enroll in the study.

This will be an exploratory study, insofar as eligible and consented informal caregivers will complete a baseline data collection session for participant characterization; they will also have the opportunity to test the ElliQ messaging function for the 2 months while their study partner (i.e., the ElliQ user) tests the ElliQ system. Informal caregivers will have the opportunity to discuss their ElliQ experience, caregiving experience, and their perception of the impacts the ElliQ system and messaging function had on their study partner's social engagement, loneliness, access to technology, and use of different communication methods (e.g., online, in-person, over the phone, etc.). An audio-recorded focus group or interview (where field notes will be taken) will be held with informal caregivers at the end of the ElliQ users' 2-month test/use period (i.e., on or around week 9 for caregivers of users in the intervention group, or on or around week 18 for caregivers of users in the waitlist control group).

The teams at Baycrest and JSLG will follow a similar protocol (for both users and informal caregivers) and will submit applications for ethics approval through the Baycrest Research Ethics Board and University of California, San Francisco (UCSF) Institutional Review Board and the JSLG Research Committee.

Recruitment

Users

For this study, the teams at Baycrest will be recruiting up to 50 participants and JSLG will be recruiting up to 50 participants (i.e., users) at each site, with the aim of recruiting a total of 100 participants. Participants will include residents at Baycrest or JSLG/UCSF, as well as community-dwelling older adults who live within the vicinity of Baycrest or JSLG/UCSF. Recruitment will occur on an ongoing basis at both Baycrest and JSLG.

Recruitment venues

1. San Francisco, JSLG in Partnership with UCSF (n=50)
2. Baycrest (n=50)

Participant consent will adopt the tenets of the Partnership of Consent Protocol, whereby the prospective participant (or their substitute decision maker, if applicable) will review the consent form with research staff. Consent will be obtained from the prospective participant (or their SDM), if they are able to provide it and can answer the teach-back questions.

Informal Caregivers

Study participants (users) will be asked by the research staff if they have an informal caregiver (e.g., a family member or friend who provides care for them) who might be interested in taking part in the study as well. Those participants who indicate that they do have an informal caregiver who might be interested will be provided with the research staff's contact information to share with their informal caregiver. Interested caregivers who contact the research staff will be provided with more information about the study either over the phone, in person, or over email. Users who do not have informal caregivers can still take part in the study and will not have access to the messaging function.

ELIGIBILITY:
Inclusion Criteria (Users):

* Older adults aged ≥70 years old and living alone
* Has minimal exposure to technology on a daily basis
* Residents of Baycrest or JSLG/UCSF, or community-dwelling older adults who live near Baycrest or JSLG/UCSF
* Agrees to allow the ElliQ setup team (a member of Baycrest or JSLG/UCSF and Intuition Robotics) to come to their home to install the ElliQ system and to provide training on how to use the system
* Agrees to have the ElliQ setup team test their existing Wi-Fi in their home or agrees to allow for installation of Wi-Fi in their home for the duration of the study (at no cost to the participant)
* Is able to speak clearly and be understood, as exemplified by an app such as Siri/Google speech recognition
* Is able to hear a finger rub with hearing aids in, if applicable
* Is able to read visual content on a screen

Exclusion Criteria (Users):

* Is unable to communicate in oral English
* Is unable to read visual content on a screen
* Has a history or current diagnosis of major psychiatric conditions, excluding depression
* Has sensory impairments (e.g., severe auditory or visual impairments) that would impede an individual's ability to interact with the ElliQ system, which features voice-activated technology and the presentation of content on a screen
* Has a Mini-Mental State Examination (MMSE) score <18
* Is currently enrolled in another study

Inclusion Criteria (Informal Caregivers):

* Is an informal caregiver (e.g., a family member, friend, etc.) of an ElliQ study participant
* Lives separately (in a different home) from their study partner (i.e., the ElliQ participant)
* Has access to an Android Smartphone or iPhone running iOS v. 10 or above through which to access Twilio Messenger
* Is willing and able to use Twilio Messenger to access the ElliQ messaging function
* Understands and abides by the terms and conditions of the messaging app (i.e., Twilio messenger) that links to the ElliQ system
* Is able to speak clearly and in oral English
* Able to hear audio and see and read content on a screen

Exclusion Criteria (Caregivers):

* Individuals who are not an informal caregiver to an ElliQ study participant
* Lives in the same home as the ElliQ study participant
* Does not have access to an Android Smartphone or iPhone running iOS v. 10 or above through which to access Twilio Messenger
* Is unable or unwilling to use Twilio Messenger to access the ElliQ messaging function
* Refuses to abide by the terms and conditions of Twilio Messenger
* Is unable to speak or read in English
* Is unable to hear audio or see/read content on a screen

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
University of California, Los Angeles Loneliness (UCLA) V3 Scale - Change is Being Assessed | Time 1 (baseline, week 0), Time 2 (follow-up 1, week 9), Time 3 (follow-up 2, week 18)
  The UCLA Loneliness V3 scale is a 20-item scale measuring loneliness and social isolation; it has been validated in older adult populations. For this scale, 11 items are worded negatively to indicate loneliness, while 9 are worded positively (and are reverse scored) to indicate social connectedness. Participants are asked to rate their responses on a 4-point scale, with responses ranging from 1 ("never") to 4 ("often"). The individual items are then tallied and a total score is calculated (range: 20-80). Higher scores indicate higher levels of loneliness. As the primary outcome for this study, the investigators are exploring the impacts of the social robot on participants' self-rated loneliness/social connectedness. This measure is being collected at multiple time points to evaluate whether there is a change observed across loneliness over time.

OTHER OUTCOMES:
Computer Proficiency Questionnaire | Time 1 (baseline, week 0), Time 2 (follow-up 1, week 9), Time 3 (follow-up 2, week 18)
  A questionnaire assessing individuals' proficiency with technology use; this measure has been validated in older adult populations
ElliQ Companionship Questionnaire | Time 2 (follow-up 1, week 9), Time 3 (follow-up 2, week 18)
  A novel questionnaire assessing participants' experiences with the social robot
Caregiver Status | Time 1 (baseline, week 0), Time 2 (follow-up 1, week 9), Time 3 (follow-up 2, week 18)
  A novel questionnaire assessing participants' access to caregiver support
Duke's Social Support Index (DSSI) | Time 1 (baseline, week 0), Time 2 (follow-up 1, week 9), Time 3 (follow-up 2, week 18)
  The DSSI is an 11-question survey measuring social engagement and social connectedness; this measure has been validated in older adult populations. The DSSI is measured by summing the total score of 10 of 11 items. Scores can range from 11-33, with higher scores indicating access to more social support. The DSSI also includes subscales, with items 1-4 measuring social interaction (range: 4-12; higher scores indicate greater social interaction), and items 5-11 measuring subjective social support (range: 7-21; higher scores indicate greater social support). Changes in the total score and across subscales will be evaluated as part of this study.
Old People's Quality of Life-Brief (OPQOL-Brief) | Time 1 (baseline, week 0), Time 2 (follow-up 1, week 9), Time 3 (follow-up 2, week 18)
  The OPQOL-Brief questionnaire assesses quality of life in older adults. This 13-item questionnaire examines respondents' quality of life across different domains (home/neighbourhood, leisure activities, social activities, life satisfaction, control in life, and well-being). For each item, respondents indicate the extent they agree or disagree with a given statement, where responses range from 1 ("Strongly disagree") to 5 ("Strongly agree)". Scores can range from 13-65; higher scores indicate higher quality of life ratings. Changes in the total score will be evaluated.
Brief Mood Introspection Scale (BMIS) | Time 1 (baseline, week 0), Time 2 (follow-up 1, week 9), Time 3 (follow-up 2, week 18)
  The BMIS is a 16-item scale exploring participants' mood at a given point in time; this scale has been validated in older adult populations. Participants are presented with different mood-related adjectives (e.g., "lively", "fed up") and are asked to rate the extent to which each describes their present mood. Responses range from 1 ("definitely do not feel") to 4 ("definitely feel"), and the total score ranges from 16-64. There is also one question assessing participants' overall mood, which ranges from -10 ("very unpleasant") to 10 ("very pleasant"). Subscales include "overall pleasant-unpleasant mood", "arousal-calm mood", "positive-tired mood", and "negative-calm mood". The total score and subscale scores are summed, and negative adjectives are reverse scored. Changes in the total score and across subscales will be evaluated as part of this study.
Visual Analog Mood Scale (VAMS) | Time 1 (baseline, week 0), Time 2 (follow-up 1, week 9), Time 3 (follow-up 2, week 18)
  The VAMS comprises a series of visual analog scales measuring mood; this measure has been validated in older adult populations. Participants are asked to indicate their current mood across a series of scales that range from 0-100. Each scale presents illustration pairs; the top illustration always represents a "neutral" emotional state relative to the bottom illustration, which represents a different mood (e.g., "Sad", "Happy"). Participants indicate their current mood, and raw scores (range: 0 ["Neutral"] to 100 [emotional state]) are noted for each illustration pair. All raw scores for each scale are transformed into T-scores. Negative moods: T-scores less than or equal to 59 are within normal limits, 60-69 represent borderline T-scores, and scores greater than or equal to 70 are abnormal. Positive moods: scores greater than or equal to 41 are within normal limits, 31-40 are borderline, and at or below 30 are abnormal. Changes in the total score will be evaluated.
Personal Health Questionnaire-8 (PHQ-8) | Time 1 (baseline, week 0), Time 2 (follow-up 1, week 9), Time 3 (follow-up 2, week 18)
  The Personal Health Questionnaire (PHQ)-8 is an 8-item questionnaire assessing the frequency of depressive-type symptoms; this measure has been validated in older adult populations. Respondents are asked to indicate how often they were bothered by various experiences (e.g., "Little interest or pleasure in doing things") over the course of the past two weeks. The scale for each item ranges from 0 ("Not at all") to 3 ("Nearly every day"). The total score is the sum of 8 items. Scores 1-9 are within normal limits, 10-19 indicate suspicion of major depression, and 20+ indicate suspicion for severe major depression. Changes in the total score will be evaluated as part of this study.
Focus group/interview guide - Users | Post-intervention (follow-up 1, week 9 for the group receiving the intervention first; follow-up 2, week 18 for the group receiving the intervention second)
  A focus group or interview guide that was created to examine users' experiences with and impressions of the ElliQ system
Focus group/interview guide - Caregivers | Post-intervention (follow-up 1, week 9 for the group receiving the intervention first; follow-up 2, week 18 for the group receiving the intervention second)
  A focus group or interview guide that was created to examine caregivers' experiences with and impressions of the ElliQ system and the associated messaging function

CONTACTS AND LOCATIONS:
Overall Officials: Allison B Sekuler, PhD, Principal Investigator — Baycrest
Locations (2):
- Jewish Senior Living Group, San Francisco, California, United States
- Baycrest, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batchelor-Aselage M, Amella E, Zapka J, Mueller M, Beck C. Research with dementia patients in the nursing home setting: a protocol for informed consent and assent. IRB. 2014 Mar-Apr;36(2):14-20. No abstract available. PMID 24783377
- [Background] Hastings SN, George LK, Fillenbaum GG, Park RS, Burchett BM, Schmader KE. Does lack of social support lead to more ED visits for older adults? Am J Emerg Med. 2008 May;26(4):454-61. doi: 10.1016/j.ajem.2007.07.005. PMID 18410815
- [Background] Smith JM. Toward a better understanding of loneliness in community-dwelling older adults. J Psychol. 2012 May-Jun;146(3):293-311. doi: 10.1080/00223980.2011.602132. PMID 22574422
- [Background] Mayer JD, Gaschke YN. The experience and meta-experience of mood. J Pers Soc Psychol. 1988 Jul;55(1):102-11. doi: 10.1037//0022-3514.55.1.102. PMID 3418484
- [Background] Machado L, Thompson LM, Brett CHR. Visual analogue mood scale scores in healthy young versus older adults. Int Psychogeriatr. 2019 Mar;31(3):417-424. doi: 10.1017/S1041610218000996. Epub 2018 Jul 11. PMID 29991360
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Bowling A, Stenner P. Which measure of quality of life performs best in older age? A comparison of the OPQOL, CASP-19 and WHOQOL-OLD. J Epidemiol Community Health. 2011 Mar;65(3):273-80. doi: 10.1136/jech.2009.087668. Epub 2010 Aug 18. PMID 20719807
- [Background] Bichescu-Burian D, Cerisier C, Czekaj A, Grempler J, Hund S, Jaeger S, Schmid P, Weithmann G, Steinert T. [Patients with ICD-10 disorders F3 and F4 in psychiatric and psychosomatic in-patient units - who is treated where? : Allocation features from the PfAD study]. Nervenarzt. 2017 Jan;88(1):61-69. doi: 10.1007/s00115-015-0058-9. German. PMID 26842897
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Boot WR, Charness N, Czaja SJ, Sharit J, Rogers WA, Fisk AD, Mitzner T, Lee CC, Nair S. Computer proficiency questionnaire: assessing low and high computer proficient seniors. Gerontologist. 2015 Jun;55(3):404-11. doi: 10.1093/geront/gnt117. Epub 2013 Oct 9. PMID 24107443
- [Background] Kopecek M, Bezdicek O, Sulc Z, Lukavsky J, Stepankova H. Montreal Cognitive Assessment and Mini-Mental State Examination reliable change indices in healthy older adults. Int J Geriatr Psychiatry. 2017 Aug;32(8):868-875. doi: 10.1002/gps.4539. Epub 2016 Jun 29. PMID 27352935
- [Background] Koskas P, Henry-Feugeas MC, Feugeas JP, Poissonnet A, Pons-Peyneau C, Wolmark Y, Drunat O. The Lawton Instrumental Activities Daily Living/Activities Daily Living Scales: A Sensitive Test to Alzheimer Disease in Community-Dwelling Elderly People? J Geriatr Psychiatry Neurol. 2014 Jun;27(2):85-93. doi: 10.1177/0891988714522694. Epub 2014 Feb 26. PMID 24578460
- [Background] Jakobsson U, Westergren A, Lindskov S, Hagell P. Construct validity of the SF-12 in three different samples. J Eval Clin Pract. 2012 Jun;18(3):560-6. doi: 10.1111/j.1365-2753.2010.01623.x. Epub 2011 Jan 6. PMID 21210901
- [Background] Poscia A, Stojanovic J, La Milia DI, Duplaga M, Grysztar M, Moscato U, Onder G, Collamati A, Ricciardi W, Magnavita N. Interventions targeting loneliness and social isolation among the older people: An update systematic review. Exp Gerontol. 2018 Feb;102:133-144. doi: 10.1016/j.exger.2017.11.017. Epub 2017 Dec 2. PMID 29199121
- [Background] Jones RB, Ashurst EJ, Atkey J, Duffy B. Older people going online: its value and before-after evaluation of volunteer support. J Med Internet Res. 2015 May 18;17(5):e122. doi: 10.2196/jmir.3943. PMID 25986724
- [Background] Robinson H, Macdonald B, Kerse N, Broadbent E. The psychosocial effects of a companion robot: a randomized controlled trial. J Am Med Dir Assoc. 2013 Sep;14(9):661-7. doi: 10.1016/j.jamda.2013.02.007. Epub 2013 Mar 30. PMID 23545466
- [Background] Boss L, Kang DH, Branson S. Loneliness and cognitive function in the older adult: a systematic review. Int Psychogeriatr. 2015 Apr;27(4):541-53. doi: 10.1017/S1041610214002749. Epub 2015 Jan 2. PMID 25554219
- See also: Statistics Canada. Canada Year Book. 2011. — https://www150.statcan.gc.ca/n1/en/pub/11-402-x/2011000/pdf/seniors-aines-eng.pdf?st=3WtalrlC

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT03972787/Prot_SAP_000.pdf